CLINICAL TRIAL: NCT04866667
Title: Screening and Intervention of Arteriosclerotic Cardiovascular Disease in Type 2 Diabetes in Zhejiang Province
Brief Title: Observational Study of ASCVD Risks of Type 2 Diabetes in East China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Zhejiang Provence Preventive Medicine Association (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); Affiliated Cixi Hospital of Wenzhou Medical University (Other); Putuo People's Hospital (Unknown); The Second People's Hospital of Yuhuan (Unknown); Affiliated Wenling Hospital of Wenzhou Medical University (Other); ShuGuang Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Nanxun People's Hospital (Unknown); The First People's Hospital of Huzhou (Other); Lishui Hospital of TCM (Unknown); Hangzhou hospital of Chinese Traditional Medicine (Unknown); Zhejiang Greentown Cardiovascular Hospital (Other); Red Cross Hospital, Hangzhou, China (Other); The Second School of Medicine，WMU (Unknown); The First People's Hospital of Xiaoshan (Unknown); Zhejiang Hospital (Other); Yiwu Central Hospital (Other); Quzhou Hospital (Unknown); Jinhua Hospital of TCM (Unknown); Shaoxing Central Hospital (Other); Shaoxinig Second Hospital (Unknown); Huamei hospital, University of Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Xiao Ye, MD, Director Assistant, Zhejiang Provincial People's Hospital
Other Study IDs: zjPPHNFM001
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus; Arteriosclerotic Cardiovascular Disease; Liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- antidiabetic drugs including GLP-1 RAs: Apply Type 2 Diabetes mellitus patients with high risk of ASCVD with antidiabetic drugs including GLP-1 RAs
- antidiabetic drugs not including GLP-1 RAs: Apply Type 2 Diabetes mellitus patients with high risk of ASCVD with antidiabetic drugs not including GLP-1 RAs，such as metformin，insulin

SUMMARY:
The aim of this study is to screen patients with type 2 diabetes with high risk of cardiovascular disease, and intervene with or without Glucagon like peptide-1 receptor agonists.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c ≥7.0%
* Prior CVD cohort: age ≥50 and ≥1 of the following criteria.

  * Prior MI
  * Prior stroke or TIA
  * Prior coronary, carotid or peripheral arterial revascularization
  * N50% stenosis of coronary, carotid, or lower extremity arteries
  * History of symptomatic CHD documented by Positive exercise stress test or any cardiac imaging or Unstable angina with ECG changes
  * Asymptomatic cardiac ischemia Documented by positive nuclear imaging test, exercise test or dobutamine stress echo
  * Chronic heart failure NYHA class II-III
  * Chronic renal failure, eGFR <60 mL/min per 1.73m2 MDRD eGFR <60 mL/min per Cockcroft-Gault formula
* No Prior CVD group: Age ≥60 y and ≥1 of the following criteria.

  * Microalbuminuria or proteinuria
  * Hypertension and left ventricular hypertrophy by ECG or imaging
  * Left ventricular systolic or diastolic dysfunction by imaging
  * Ankle-brachial index b0.9

Exclusion Criteria:

* Type 1 diabetes
* other type diabetes
* Calcitonin ≥50 ng/L
* Use of a GLP-1 receptor agonist (exenatide, liraglutide or other) or pramlintide or any DPP-4 inhibitor within the 3 months prior to screening
* Use of insulin other than human NPH insulin or long-acting insulin analogue or premixed insulin within 3 months prior to screening. Shortterm use of other insulin during this period in connection with intercurrent illness is allowed, at Investigators discretion
* Acute decompensation of glycemic control
* An acute coronary or cerebrovascular event in the previous 14 d
* Currently planned coronary, carotid, or peripheral artery revascularization
* Chronic heart failure (NYHA class IV)
* Current continuous renal replacement therapy
* End-stage liver disease
* History of solid organ transplant or awaiting solid organ transplant
* Malignant neoplasm
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients over 18 years old with high risks of atherosclerotic cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
New-onset cardiovascular events | maximum 2 years
  Composite of angina pectoris, stroke, myocardial infarction, atherosclerotic plaque，unplanned rehospitalization, stent thrombosis, incidence of cardiac death in the duration of follow-up

SECONDARY OUTCOMES:
Blood glucose control | maximum 2 years
  Change of fasting and postprandial blood glucose in the duration of follow-up
Lipid levels | maximum 2 years
  Change of lipid levels（Total cholesterol, Total triglycerides, low density lipoprotein，high density lipoprotein） in the duration of follow-up
Blood pressure level | maximum 2 years
  Change of blood pressure（mmHg） in the duration of follow-up
Body weight | maximum 2 years
  Change of body weight(kg) in the duration of follow-up
Fat Distribution Indicators | maximum 2 years
  Change of abdomen circumference（cm） in the duration of follow-up
Fat Distribution Indicators | maximum 2 years
  Change of waist circumference（cm） in the duration of follow-up
Microvascular complications | maximum 2 years
  Microvascular complications（such as Diabetic retinopathy，Diabetic nephropathy） in the duration of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Wu, MD, Principal Investigator — Department of Endocriology, Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No
No plan to share data